CLINICAL TRIAL: NCT00612625
Title: Near Normalisation of Blood Glucose Improves the Potentiating Effect of GLP-1 on Glucose Induced Insulin Secretion in Patients With Type 2 Diabetes
Brief Title: Near Normalisation of BG Improves the Potentiating Effect of GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Patricia Verdugo Højberg, MD, PHD, Patricia Verdugo Højberg
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: KF 01 - 198/03; KA 01 - 198/03
Record Dates: First submitted 2008-01-16; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP-1 (Experimental): A graded glucose infusion with an infusion of GLP-1 (1½ pmol/kg/min)
  Interventions: Drug: glucagon-like peptide-1
- Saline (Experimental): A graded glucose infusion together with a continuous infusion of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: glucagon-like peptide-1 — continuous infusion of GLP-1 (1½ pmol/kg/min)
  Arms: GLP-1
Drug: Saline — continuous infusion of saline
  Arms: Saline

SUMMARY:
The ability of glucagon-like peptide 1 to enhance beta-cell responsiveness to I.v. glucose is impaired in patients with type 2 diabetes mellitus compared with healthy individuals. We investigated whether 4 weeks of near-normalisation og blood glucose improves the potentiation of glucose-stimulated insulin secretion by GLP-1

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Type 2 diabetes diagnosed after 30 years of age
* BMI > 25

Exclusion Criteria:

* Severe complications to diabetes
* Abnormal liver og kidney function
* Haemoglobin below the lower limit
* Macroalbuminuria
* Systemic disease
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2004-02; Primary Completion 2004-07 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
insulin secretion rate (ISR) were derived by deconvolution of c-peptide. ISR is expressed as pmol/kg/min | 180 minutes

SECONDARY OUTCOMES:
The calculated ISR values was plotted against the ambient plasma glucose. The slopes of this linear relationships were calculated by cross-correlation analysis and is and estimation of beta-cell responsiveness (pmol/kg/min)/mmol/l | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Patricia V Højberg, MD, PHD, Principal Investigator — University Hospital Hvidovre
Locations (1):
- Dept. of Endocrinology, Hvidovre Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Hojberg PV, Zander M, Vilsboll T, Knop FK, Krarup T, Volund A, Holst JJ, Madsbad S. Near normalisation of blood glucose improves the potentiating effect of GLP-1 on glucose-induced insulin secretion in patients with type 2 diabetes. Diabetologia. 2008 Apr;51(4):632-40. doi: 10.1007/s00125-008-0943-x. Epub 2008 Feb 22. PMID 18292985